CLINICAL TRIAL: NCT04426617
Title: Comparison Between Fentanyl And Midazolam As Additives To Bupivacaine In Ultrasound Guided Transversus Abdominis Plane Block in Patients Undergoing Abdominal Surgeries; A Randomized Controlled Study
Brief Title: Fentanyl Versus Midazolam As Additives To Bupivacaine In Ultrasound Guided Transversus Abdominis Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bassant M. Abdelhamid (Other)
Responsible Party: Sponsor-Investigator, Bassant M. Abdelhamid, Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-258-2019
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- fentanyle (Experimental): : patients will receive US guided unilateral Transversus abdominis plane block (25 ml bupivacaine 0.25% & fentanyl).
  Interventions: Procedure: Ultrasound Guided Transversus Abdominis Plane Block
- Midazolam (Experimental): patients will receive us guided unilateral Transversus abdominis plane block (25 ml bupivacaine 0.25% & midazolam).
  Interventions: Procedure: Ultrasound Guided Transversus Abdominis Plane Block
- control (Placebo Comparator): patients will receive us guided unilateral Transversus abdominis plane block (25 ml bupivacaine 0.25%).
  Interventions: Procedure: Ultrasound Guided Transversus Abdominis Plane Block

INTERVENTIONS:
Procedure: Ultrasound Guided Transversus Abdominis Plane Block — The patient will lie in the supine position. The transducer will be placed in the axial plane on the mid-axillary. transversus abdominis muscle will be visualized. A skin wheel using 3 ml of lidocaine 1 % is made 2 to 3 cm medial to the medial aspect of the transducer and the 22 gauge is inserted in-plane pointing laterally. Then Injection of local anaesthetic mixure in the right plane.

SUMMARY:
Pain triggers a complex biochemical and physiological stress response leading to impairment of pulmonary, immunological and metabolic functions.

The Transversus Abdominis Plane (TAP) block, is a regional anaesthesia technique used for various surgeries through the lower to mid-abdominal wall.The addition of fentanyl to the local anaesthetic in ultrasound-guided TAP block prolongs the analgesia, lowers postoperative pain, and decreases the opioid consumption. Adding midazolam as a bupivacaine adjuvant for TAP block reduces the 24-h morphine consumption extends the postoperative analgesia duration. The aim of the work is to study the effect of the addition fentanyl and midazolam on the onset, duration of the analgesic effect of Tap block intraoperative fentanyl consumption, Time for first rescue Analgesia.

in patients undergoing simple unilateral abdominal surgeries.

DETAILED DESCRIPTION:
Informed written consent will be obtained from study participants or their legally authorized representative. This is a randomized controlled double blinded study; patients will be enrolled in the study and will be randomized and equally divided into three groups:

Group A: (TAP block with 20 ml of bupivacaine 0.25% and 50 μ g of fentanyl) Group B: (TAP block with 20 ml bupivacaine 0.25% and 50 μ g /kg midazolam) Group C: (TAP block with 20 ml bupivacaine 0.25% only). Induction of general anaesthesia will be performed using a regimen of IV 1 μ g/kg fentanyl and Propofol IV 2 mg /kg. Tracheal intubation will be facilitated using 0.5 mg/kg IV of atracurium.

Maintenance of Anaesthesia:

Anaesthesia will be maintained with inhaled sevoflurane with MAC 2% in oxygen enriched air (FiO2=0.5) and top up doses of Atracurium (0.1 mg/kg) IV will be administered every 30 minutes.

Ringer acetate will be infused to replace their fluid deficit, maintenance and losses, and the patients will be mechanically ventilated using the appropriate setting that will keep the end-tidal CO2 at 30-35mmHg.

One reading of mean arterial pressure (MAP) and heart rate (HR) will be taken 1 minute before induction of general anaesthesia (a baseline reading), 1 minute before surgical incision and at 15-minute intervals intra operatively.

Lack of inadequate intraoperative analgesia, as defined by an increase in pulse rate, sweating, and tearing (PRST) score >2 or an increase of mean arterial blood pressure (MAP) >20% of baseline (8) was treated by additional rescue IV fentanyl 1-2 mcg/kg IV bolus.

Hypotension will be treated with 0.9% normal saline and/or 5mg ephedrine in incremental doses to maintain mean blood pressure above 70 mmHg.

The residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), and extubation will be performed after complete recovery of the airway reflexes.

The patient will be transferred to the post-anaesthesia care unit (PACU) where the MAP and HR will be recorded immediately upon arrival.

Side effects such as local anaesthetic toxicity, postoperative nausea and vomiting (PONV), respiratory depression (respiratory rate <10/minute) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Physical status ASA I and ASA ll.
* Age ≥ 18 and ≤ 65 Years.
* Body mass index (BMI): ≥ 20 kg/m2 and ≤ 35 kg/m2.
* Patients undergoing Abdominal Surgeries.
* Patient is able to provide a written informed consent.

Exclusion Criteria:

* Known sensitivity to local anaesthetics.
* Significant liver or renal insufficiency.
* Contraindication to regional anaesthesia e.g. local - sepsis, pre-existing peripheral neuropathies and coagulopathy.
* Patient refusal.
* Failed Block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Onset of the Analgesic effect of TAP block with different additives | 30 minutes
  The patient will be asked to register a prick respectively on the upper extremity. Sensory change will then be assessed in the mid-clavicular line, starting above dermatome T4 moving caudally to dermatome L4.

SECONDARY OUTCOMES:
Dose of intra-Operative fentanyl consumption | 2 hours
  Lack of inadequate intraoperative analgesia, as defined by an increase in pulse rate, sweating, and tearing (PRST) score >2 or an increase of mean arterial blood pressure (MAP) >20% of baseline was treated by additional rescue IV fentanyl 1-2 mcg/kg IV bolus.
Block related complications | 24 hours
  haematoma, neurological complications
Time of first analgesic request | 24 hours
  visual analogue scale equals or more than 4
Incidence of postoperative nausea and vomiting | 24 hours postoperative
  will be assessed using by yes/ no scale

CONTACTS AND LOCATIONS:
Overall Officials: yahia hammad, M.D., Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nehra P, Oza V, Parmar V, Fumakiya P. Effect of Addition of Fentanyl and Clonidine to Local Anesthetic Solution in Peribulbar Block. J Pharmacol Pharmacother. 2017 Jan-Mar;8(1):3-7. doi: 10.4103/jpp.JPP_109_16. PMID 28405129
- [Background] Carney J, Finnerty O, Rauf J, Bergin D, Laffey JG, Mc Donnell JG. Studies on the spread of local anaesthetic solution in transversus abdominis plane blocks. Anaesthesia. 2011 Nov;66(11):1023-30. doi: 10.1111/j.1365-2044.2011.06855.x. Epub 2011 Aug 18. PMID 21851346
- [Result] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150